



# **Nurse Participant Information and Consent Form**

1. Duration of urinary catheterization following cesarean deliveries under neuraxial anesthesia: a prospective cohort study (DUCC Study)

2. Study personnel

Principal Investigator: Anton Chau, MD MMSC FRCPC

Department of Anesthesia BC Women's Hospital Phone: 604-875-2158

Lead Investigator: Aislynn Sharrock, BA (Hons.)

Department of Anesthesia BC Women's Hospital Phone: 604-875-2158

**Co-Investigators:** Marianne Vidler, PhD

Juliana Barrera, MD MSc FRCPC

Neither the Principal Investigator nor the Co-Investigators have received financial compensation from any sponsor for the work required in doing this clinical research.

#### **Study Contact Number:**

- During Office Hours (Mon-Fri; 8:30am-4:30pm): 604-875-2158, ask the Department of Anesthesia administrative assistant to page one of the study investigators.
- Outside Office Hours: 604-875-2161, ask the operator to page the Anesthesiologist on Call.

#### 3. Invitation

You are being invited to take part in this research study because you are a nurse taking care of a patient who underwent a cesarean delivery under neuraxial anesthesia at BC Women's Hospital.

# 4. Your participation is voluntary

Your participation is voluntary. You have the right to refuse to participate in this study. If you decide to participate, you may still choose to withdraw from the study at any time without any negative consequences.





Please review the consent document carefully when deciding whether or not you wish to be part of the research and sign this consent only if you accept being a research participant.

# 5. Who is conducting this study?

This study is being conducted by the Department of Anesthesia at BC Women's Hospital in Vancouver, British Columbia. The Principal Investigator is Dr. Anton Chau, and the study co-investigators are Ms. Aislynn Sharrock, Dr. Marianne Vidler, and Dr. Juliana Barrera.

This study is not receiving funds from any external agency or sponsor and none of the study researchers have any conflicts of interest to disclose.

# 6. Background

In cesarean deliveries, urinary catheters are often used to help empty the bladder while patients have limited mobility. These catheters typically stay in during early recovery because certain pain medications can make it hard for patients to urinate. Recently, the Society of Obstetric Anesthesia and Perinatology (SOAP) recommended removing catheters within 6–12 hours after delivery to aid recovery. However, at BC Women's Hospital, a review found that catheters stayed in for an average of 19 to 19.4 hours, even when patients were mobile.

Leaving catheters in too long can increase the risk of urinary tract infections (UTIs), pain, and urination issues, which can delay recovery and extend hospital stays. An internal review showed that factors like patient anxiety may affect when catheters are removed. Postpartum anxiety affects around 9.9% to 20.7% of new mothers in the first year and is an important factor in recovery after a cesarean delivery.

#### 7. What is the purpose of the study?

The main goal of this study is to see if there is a link between duration of catheter and patient's anxiety level measured from a questionnaire. In addition to asking patients to fill in the questionnaire, we want to look at nursing factors that could influence how long urinary catheters stay in patients.

# 8. Who can participate in this study?

You may be able to participate in this study if you are a nurse taking care of a patient who underwent a cesarean delivery under neuraxial anesthesia at BC Women's Hospital.

#### 9. Who should not participate in this study?

You will not be eligible to participate in this study if you refuse to participate and if you are taking care of a patient that delivered by cesarean section under general anesthesia or other non-cesarean surgeries.





# 10. What does the study involve?

# • If You Decide to Join This Study: Specific Procedures

If you agree to take part in this study, the procedures and visits you can expect will include the following:

# • Study Visit

You will be approached by research staff if you are taking care of a postpartum patient who underwent a cesarean delivery and is recovering in a postpartum ward. At an appropriate time, you will be asked to answer questions regarding your assessment of your patient's urinary catheter. At the time research staff approaches, your patient will either already have their catheter removed by you or they will still have their catheter in, and you are the nurse who is taking care of this patient. You will be asked to answer a few questions about what factors influenced the duration of the urinary catheter being left in based on your assessment of the patient. The questionnaire will be anonymized and no personal or identifying information from you will be collected. This questionnaire should only take 2 minutes to answer.

# Communication of patient pain and anxiety scores

As part of this study, we will also be asking patients to fill out a questionnaire about their current postpartum pain and current feelings of anxiety. If research staff observes findings through the patient's data collection form that could be of potential clinical relevance (e.g., high pain or anxiety scores), the patient will be asked if they would like the research staff to relay this information to their circle of care. If the patient gives us permission, research staff will contact their most responsible physician (MRP) and/or nursing staff to relay this information on their data collection form. In these instances, you may be approached by research staff for the purpose of relaying the information to you. The research staff will not be interpreting the findings or offering clinical referrals to the patient participants.

## 11. What are the possible harms and discomforts?

There are no risks for joining this study.

# 12. What are the potential benefits of participating?

There may not be direct benefit to you from taking part in this study. We hope that the information learned from this study can be used in the future to improve patient's recovery after a cesarean delivery under neuraxial anesthesia.

#### 13. After the study is finished





We believe that this study will take about 9 months to complete. If you are interested in knowing the results of the study, please contact the Department of Anesthesia at 604-875-2158 and one of the study investigators will contact you.

# 14. What happens if I decide to withdraw my consent to participate?

You may withdraw from this study at any time without giving reasons. If you choose to enter the study and then decide to withdraw at a later time, you have the right to request the withdrawal of your information collected during the study. This request will be respected to the extent possible. Please note however that there may be exceptions where the data will not be able to be withdrawn for example where the data is no longer identifiable (meaning it cannot be linked in any way back to your identity) or where the data has been merged with other data. If you would like to request the withdrawal of your data, please let the principal investigator of the study know.

# 15. How will my taking part in this study be kept confidential?

Your confidentiality will be respected. However, research records and health or other source records identifying you may be inspected in the presence of the Investigator or designate and by representatives of UBC Children's and Women's Research Ethics Board, for the purpose of monitoring the research. No information or records that disclose your identity will be published without your consent, nor will any information or records that disclose your identity be removed or released without your consent unless required by law.

Because this study is primarily focused on data from patients, no identifiable information related to you will be included in our data collection. The questionnaire you fill out will be paired with the patient's data. The patient will be assigned a unique study number as a participant in this study. Only this number will be used on any research-related information collected about the patient and their paired questionnaire filled out by you during the course of this study.

Your rights to privacy are legally protected by federal and provincial laws that require safeguards to ensure that your privacy is respected. You also have the legal right of access to the information about you, if need be, an opportunity to correct any errors in this information. Further details about these laws are available on request to the study team.

#### 16. Future Use of Data

The prospective cohort study will be published in a medical journal and presented at conferences so that we can disseminate the findings within the medical community. It is our hope that this study will catalyze ongoing research to further enhance postpartum recovery following cesarean delivery under neuraxial anesthesia.





We only anticipate the Primary Investigator and study team members to have access to the data for the purposes of completing the objectives of this study.

# 17. What happens if something goes wrong?

By signing this form, you do not give up any of your legal rights and you do not release the principal investigator, participating institutions, or anyone else from their legal and professional duties.

#### 18. What will the study cost me?

You will not incur any personal expenses as a result of participation in this study, nor will you be paid for participating.

# 19. If I have questions about the study procedures during my participation, who should I speak to?

If you have any questions or desire further information about this study before or during participation you can contact Aislynn Sharrock (Co-Investigator) or Anton Chau (Principal Investigator) at 604-875-2158. You can also reach the anesthesiologist on call at any time at 604-875-2161 (24-hour paging number).

# 20. Who do I contact if I have any questions or concerns about my rights as a participant?

If you have any concerns or complaints about your rights as a research participant and/or your experiences while participating in this study and/or have any concerns or complaints related to privacy, contact the Research Participant Complaint Line in the University of British Columbia Office of Research Ethics by e-mail at RSIL@ors.ubc.ca or by phone at 604-822-8598 (Toll Free: 1-877-822-8598.) Please reference the study number (H24-03410) when contacting the Complaint Line so the staff can better assist you.





#### 21. **Future Contact**

| • | to be contacted once the study in the study is siving a copy of the journal article. | * | |
|---|---|---|---|
| □ Yes □ No | Name: | Email Address: | |
| Are you intereste | ed in learning about other studio | es conducted by Dr. Anton Ch | nau in the future? |
| □ Yes □ No | Name: | Email Address: | |
| Note that for any | future studies, a separate cons | ent form will be provided to y | ou for review. |





# 22. Signatures

Duration of urinary catheterization following cesarean deliveries under neuraxial anesthesia: a prospective cohort study (DUCC Study)

#### **Participant Consent**

My signature on this consent form means:

- I have read and understood the information in this consent form.
- I have been able to ask questions and have had satisfactory responses to my questions.
- I understand that my participation in this study is voluntary.
- I understand that I am completely free at any time to refuse to participate or to withdraw from this study at any time.
- I understand that I am not waiving any of my legal rights as a result of signing this consent form.
- I understand that there is no guarantee that this study will provide any benefits to me.

| I will receive a signed and dat I consent to participate in this | * • | form for my own | records. |
|---|---|---|---|
| Participant's Signature | Printed name | ; | Date |
| Signature of Person Obtaining Consent | Printed name | Study Role | Date |